CLINICAL TRIAL: NCT05522894
Title: A Multicenter, Phase II Clinical Study of AK104 (Anti-PD-1/CTLA-4 Bispecific Antibody) Alone or in Combination With Chemotherapy in the First-line Treatment of Advanced Esophageal Squamous Cell Carcinoma
Brief Title: AK104 Alone or in Combination With Chemotherapy in the First-line Treatment of ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Principal Investigator, Jing Huang, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3649
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Unresectable Esophageal Squamous Cell Carcinoma; Locally Advanced Esophageal Squamous Cell Carcinoma; Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): AK104 alone
  Interventions: Drug: AK104
- Cohort B (Experimental): AK104 in combination with chemotherapy
  Interventions: Drug: AK104; Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: AK104 — 10mg/kg IV every 3 weeks (Q3W)
  Other Names: Cadonilimab
Drug: Cisplatin — 75mg/m2 IV every 3 weeks (Q3W)
  Other Names: DDP
  Arms: Cohort B
Drug: Paclitaxel — 175mg/m2 IV every 3 weeks (Q3W)
  Other Names: PTX
  Arms: Cohort B

SUMMARY:
This is a two-arm, open, multicenter clinical study to evaluate the efficacy and safety of AK104 alone or in combination with cisplatin and paclitaxel in the treatment of advanced esophageal squamous carcinoma without systemic therapy.

DETAILED DESCRIPTION:
During the treatment, eligible patients in cohort A with PD-L1 CPS ≥5 will receive AK104 10 mg/kg, intravenously, every 3 weeks (maximum 24 months of dosing); in cohort B, regardless of PD-L1 expression, eligible patients will receive AK104 10 mg/kg, intravenously, every 3 weeks (maximum 24 months of dosing), in combination with cisplatin (75 mg/m2) and paclitaxel (175 mg/m2), Q3W (up to 6 cycles, the specific cycles will be determined by the investigator). Thereafter, AK104 maintenance therapy will be continued until disease progression, intolerable toxicity, withdrawal of informed consent, death, or end of the study, whichever occurred first (maximum duration of treatment with AK104 should be less than 12 months). When patients with initially unresectable disease transformed into resectable, an operation can be considered and the original regimen may be used after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old, men or women are not limited
2. Histologically or cytologically confirmed as esophageal squamous cell carcinoma (including the gastroesophageal junction), (adenosquamous carcinoma with a predominantly squamous component is allowed)
3. Unresectable, locally advanced, recurrent, or metastatic esophageal squamous cell carcinoma
4. Patients who have never received systemic antitumor therapy
5. ECOG score 0-1
6. Patients who have measurable lesions that meet RECIST 1.1 criteria
7. Patients who are expected to survive more than 3 months
8. Women of childbearing age must have a negative pregnancy test (serum or urine) and voluntarily use an appropriate method of contraception
9. Patients who are voluntarily enrolled in the study and sign an informed consent form (ICF)
10. Patients who are well adherent and able to follow up the study protocol
11. Patients with normal function organs, no serious abnormalities of blood, heart, lung, liver, kidney function, and immunodeficiency diseases.
12. Patients with normal coagulation function, no active bleeding, and thrombotic disease
13. cohort A: AK104 monotherapy cohort enrolling patients with esophageal cancer tumor tissue PD-L1 CPS ≥ 5 (uniformly using Dako 22C3 antibody)

Exclusion Criteria:

1. Locally advanced esophageal cancer that can be radically resectable or potentially cured by radiotherapy
2. Other malignancies diagnosed within 5 years prior to the first administration of the study drug, except effectively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or effectively resected in situ cervical and/or breast cancer
3. Symptomatic central nervous system metastases (brain metastases confirmed stable by imaging for more than 3 months can be enrolled)
4. A serious infection (CTCAE > grade 2) such as severe pneumonia requiring hospitalization, bacteremia, or infectious comorbidities that occurred within 4 weeks prior to the first administration of the study drug; baseline chest imaging suggestive of active pulmonary inflammation with clinically relevant signs or symptoms; signs and symptoms of infection within 2 weeks prior to the first administration of study drug, or requiring oral, or intravenous antibiotic therapy. Excluding prophylactic use of antibiotics
5. Patients with previous and current interstitial pneumonia, pneumoconiosis, drug-related pneumonia, or severely impaired lung function that may interfere with the detection and management of suspected drug-related pulmonary toxicity; patients with radiation pneumonia within 6 months
6. Patients with active tuberculosis infection detected by history or CT examination, patients with a history of active tuberculosis infection within 1 year prior to enrollment, or patients with a history of active tuberculosis infection more than 1 year ago but without formal treatment
7. Patients previously treated with immune checkpoint inhibitors
8. Patients who have a congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower limit of detection of the assay) or combined hepatitis B and hepatitis C co-infection
9. Patients who have a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
10. The presence of thrombosis-type diseases or using anticoagulant drugs
11. Patients with any serious or uncontrolled systemic disease that, in the opinion of the investigator, may increase the risk associated with participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  ORR is proportion of subjects with complete response(CR) or partial response(PR), based on Response Evaluation Criteria in Solid Tumors(RECIST) v1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) is defined as the time from the first dose of investigational products until documentation of PD (as per RECIST v1.1) or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to approximately 2 years
  Overall survival (OS) is defined as the time from the first dose of investigational products until death due to any cause.
Disease control rate (DCR) | Up to approximately 2 years
  Disease control rate (DCR) is defined as the proportion of subjects achieving a best of response(BOR) of confirmed CR and PR and stable disease(SD) per RECIST v1.1.
Duration of response (DoR) | Up to approximately 2 years
  Duration of response (DoR) is defined as the period from the first documentation of confirmed response (CR or PR) to the first documentation of progressive disease(PD) (as per RECIST v1.1) or death due to any cause, whichever occurs first.
Incidence and severity of adverse events(AEs) | Up to approximately 2 years
  Incidence and severity of AEs is aim to evaluate the safety of AK104 alone or combination with chemotherapy.

OTHER OUTCOMES:
The expression of PD-L1 in tumor tissue | Up to approximately 2 years
  The expression of PD-L1 is aim to investigate the relationship between PD-L1 and anti-tumor efficacy.
The level of ctDNA in blood | Up to approximately 2 years
  The level of ctDNA is aim to investigate the relationship between ctDNA and anti-tumor efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qu W, Gao J, Zhang B, Yang M, Wang Y, Liu Y, Guo Y, Guo S, Huang J. Cadonilimab combined with taxane and cisplatin as the first-line treatment of advanced esophageal squamous cell carcinoma: an open-label, multicenter phase II trial. J Immunother Cancer. 2025 Oct 30;13(10):e012869. doi: 10.1136/jitc-2025-012869. PMID 41167638